CLINICAL TRIAL: NCT05375968
Title: Mechanism of Glucose-dependent Insulinotropic Polypeptide (GIP) on Splanchnic Venous Capacitance in Postural Tachycardia Syndrome
Brief Title: Splanchnic Venous Capacitance in Postural Tachycardia Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Cyndya Shibao, MD, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: POTS-GIP; R01HL15920301A1 (Other Grant/Funding Number: NHLBI)
Record Dates: First submitted 2022-04-19; First posted 2022-05-17 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-09

CONDITIONS: Postural Tachycardia Syndrome (POTS)
Keywords: Glucose-dependent Insulinotropic Polypeptide (GIP)
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The randomization schedule will be generated by a statistician who is not related to the study. The blinded study intervention will be infused, which medication one receives will be decided by chance, like the toss of a coin .The subjects who received saline at visit 2, will get the study drug GIP(3-30)NH2 at visit 3, and vice versa
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Changes in Splanchnic venous capacitance(SVC) before and after a 75-g oral glucose challenge (Active Comparator): To compare and measure changes in splanchnic venous capacitance and superior mesenteric arterial flow before and after a 75-g oral glucose challenge during supine and 45-degree head-up tilt positions (orthostatic challenge) for up to 3 hr. between participants with POTS (Postural Tachycardia Syndrome) and Healthy Control group
  Various GIP hormones especially GLP-1, GLP-2, glucagon, and other GI hormones before and after a 75-gram oral glucose at different timepoints through out 3 hours of the study visit
  Interventions: Diagnostic Test: Measurement of Splanchnic venous capacitance(SVC)done at Baseline and after 90 min of 75 g glucose in Healthy Controls POTS patients; Diagnostic Test: Measurement of Splanchnic venous capacitance(SVC)done at Baseline and after 90 min of 75 g glucose in Healthy Controls
- Effect of GIP antagonist GIP(3-30)NH2 Vs Saline on splanchnic venous capacitance on POTS patients (Placebo Comparator): POTS patients who participated in Aim 1, will be and randomized to either saline versus GIP antagonist (GIP(3-30)NH2) in Visit 2.
  The changes in their splanchnic venous capacitance and superior mesenteric arterial flow will be measured, before and after a 75-g oral glucose challenge during supine and 45-degree head-up tilt positions (orthostatic challenge) for up to 3 hr.
  Notably, changes in venous capacitance will be assessed using segmental impedance to measure the effect of graded positive airway pressure (CPAP) on splanchnic blood volume.
  Interventions: Drug: Compare change is SVC and SMA flow due to GIP antagonist GIP(3-30)NH2; Drug: Compare change is SVC and SMA flow due to saline

INTERVENTIONS:
Diagnostic Test: Measurement of Splanchnic venous capacitance(SVC)done at Baseline and after 90 min of 75 g glucose in Healthy Controls POTS patients — While segmental bioimpedance is monitored, continuous positive airway pressure (CPAP) will be applied sequentially at 0, 4, 8, 12, and 16 cm H2O for about 30 seconds each. This positive airway pressure will increase the intrathoracic pressure, which is transmitted to the venous circulation. Pressure (CPAP pressure, X axis) - volume (splanchnic vascular volume measured by segmental impedance and expressed as % change from baseline, Y axis) relationships are then constructed to assess for splanchnic venous capacitance
  Arms: Changes in Splanchnic venous capacitance(SVC) before and after a 75-g oral glucose challenge
Diagnostic Test: Measurement of Splanchnic venous capacitance(SVC)done at Baseline and after 90 min of 75 g glucose in Healthy Controls — While segmental bioimpedance is monitored, continuous positive airway pressure (CPAP) will be applied sequentially at 0, 4, 8, 12, and 16 cm H2O for about 30 seconds each. This positive airway pressure will increase the intrathoracic pressure, which is transmitted to the venous circulation. Pressure (CPAP pressure, X axis) - volume (splanchnic vascular volume measured by segmental impedance and expressed as % change from baseline, Y axis) relationships are then constructed to assess for splanchnic venous capacitance
  Arms: Changes in Splanchnic venous capacitance(SVC) before and after a 75-g oral glucose challenge
Drug: Compare change is SVC and SMA flow due to GIP antagonist GIP(3-30)NH2 — Participants with POTS will be randomize to either saline versus GIP(3-30)NH2 acute infusion. We will measure changes in their splanchnic venous capacitance and superior mesenteric arterial flow before and after a 75-g oral glucose challenge during supine and 45-degree head-up tilt positions (orthostatic challenge) for up to 3 hr. Notably, we will assess changes in venous capacitance using segmental impedance to measure the effect of graded positive airway pressure (CPAP) on splanchnic blood volume.
  Arms: Effect of GIP antagonist GIP(3-30)NH2 Vs Saline on splanchnic venous capacitance on POTS patients
Drug: Compare change is SVC and SMA flow due to saline — Participants with POTS will be randomize to either saline versus GIP(3-30)NH2 acute infusion. We will measure changes in their splanchnic venous capacitance and superior mesenteric arterial flow before and after a 75-g oral glucose challenge during supine and 45-degree head-up tilt positions (orthostatic challenge) for up to 3 hr. Notably, we will assess changes in venous capacitance using segmental impedance to measure the effect of graded positive airway pressure (CPAP) on splanchnic blood volume.
  Arms: Effect of GIP antagonist GIP(3-30)NH2 Vs Saline on splanchnic venous capacitance on POTS patients

SUMMARY:
Postural tachycardia syndrome (POTS) affects ≈3 million young people, characterized by chronic presyncopal symptoms characterized by dizziness, lightheadedness, and orthostatic tachycardia that occur while standing. Across-sectional survey found that 25% of these patients complains that meals rich in carbohydrates are among the factors that further exacerbate POTS's symptoms and cause a myriad of gastrointestinal symptoms.

The splanchnic circulation is the largest blood volume reservoir of the human body, storing ≈25% of the total blood volume and contributing to sudden, and large, fluctuations in the stroke volume (SV). The orthostatic changes in systemic hemodynamics are particularly magnified after meals, due to increased blood volume sequestration triggered by the release of gastrointestinal peptides with vasodilatory properties. The purpose of this study is to determine if the worsening orthostatic tachycardia and symptoms after glucose ingestion in POTS patients are due to a greater increase in splanchnic venous capacitance and excessive blood pooling on standing as compare to Healthy controls.

The study will also determine if glucose-induced GIP secretion increases splanchnic venous capacitance, orthostatic tachycardia and worsening POTS postprandial symptoms. For this purpose subjects will be further randomized to either saline versus GIP(3-30)NH2 acute infusion, to measure the changes their splanchnic venous capacitance and superior mesenteric arterial flow before and after a 75-g oral glucose challenge during supine and 45-degree head-up tilt positions (orthostatic challenge) for up to 3 hours.

DETAILED DESCRIPTION:
The Aim 1 of the study is to investigate that the worsening orthostatic tachycardia and symptoms after glucose ingestion in POTS patients are due to a greater increase in splanchnic venous capacitance and excessive blood pooling during an orthostatic challenge.

Investigators will enroll POTS patients with postprandial symptoms as cases, and age, and BMI-matched controls. The changes in their splanchnic venous capacitance and superior mesenteric arteria flow will be measured, before and after a 75-gram of oral glucose challenge, during supine and 75-degree head-up tilt positions (orthostatic challenge) for up to 3-hrs. Notably, newly developed an Innovative technique to assess venous capacitance in humans, using segmental impedance to measure the effect of graded positive airway pressure (CPAP) on splanchnic blood volume.

Rationale for Aim 1:

Several mechanisms have been associated with the pathophysiology of postprandial symptoms in POTS patients. Preliminary data showed that after a 75-g oral glucose load to POTS patients resulted in: 1) excessive increase in upright HR, which was not present in controls, 2) increased upright Heart Rate (HR), which was associated with a concomitant decrease in upright stroke volume, and 3) POTS patients had a selective increase in GIP secretion, which has vasodilatory properties in the splanchnic circulation.

There is consensus that the orthostatic tachycardia (increase upright HR), characteristic of the condition, is triggered by an exaggerated sympathetic activation, which in most cases is secondary to splanchnic venous pooling upon standing.

AIM 2 of the study, is to determine if glucose-induced GIP secretion increases splanchnic venous capacitance, orthostatic tachycardia and worsening POTS postprandial symptoms.

For this purpose, patients who participated in Aim 1, will be randomized to either saline versus GIP antagonist (GIP(3-30)NH2) acute infusion in 1:1 ratio. The changes in their splanchnic venous capacitance and superior mesenteric arterial flow will be measured, before and after a 75-g oral glucose challenge during supine and 45-degree head-up tilt positions (orthostatic challenge) for up to 3 hr. Notably, changes in venous capacitance, will be assessed, in humans using segmental impedance to measure the effect of graded positive airway pressure (CPAP) on splanchnic blood volume.

If it is assumed that higher post-glucose levels of GIP in POTS can produce a greater venodilation and a larger increase in the Y-intercept (splanchnic venous capacitance) compared to saline infusion. Then the hypothesis would be that the GIP antagonist GIP(3-30)NH2 will attenuate any increase in the Y-intercept in response to oral glucose in POTS patients

Primary endpoint: Effect of glucose on splanchnic venous capacitance in Postural Orthostatic Tachycardia Syndrome(POTS).

Secondary endpoints for aim 1 and 2 During the study, different parameters will be measured to understand the physiological cardiovascular and neuro-hormonal changes that occurred after an oral glucose intake and during orthostatic challenge in POTS patients and healthy controls. Even though these parameters will be collected during the same timepoints when the primary endpoint is collected, they are not considered study outcomes, they will inform on additional mechanisms by which glucose exert the hemodynamic and neuro-hormonal changes in POTS

Subject population: For Aim1; Total 50 participants, between age 18-50 years with BMI between 18.5 to 29.9. Out of which 25 with be participants with diagnosis of POTS and 25 heathy controls (HC).

For AIM 2 : 25 participants with diagnosis of POTS, who have completed Aim 1

Study visits: Consists of 4 visits in person:

A. Visit 0: Screening visit B. Telemedicine/phone call C. Visit 1: Baseline visit D. Visits 2 and 3 (POTS patients only)

Study procedures Visit 0/Screening visit: include EKG, urine and blood sample collection, Orthostatic Standing Test, DXA scan (dual energy X-ray absorptiometry), Measurement of blood volume using carbon monoxide rebreathing technique, Visit 1: Includes Tilt table test, Oral glucose tolerance test (OGTT), Splanchnic venous capacitance measurements.

Visit 2&3: For Aim 2: These visit will be performed under the same conditions described in Visit 1. A total of 25 POTS patients will be randomized according to a computer-generated, randomization schedule that will randomize the order of the medication order assignment (IV saline then GIP 3-30 NH2 or vice versa).The blinded study intervention will be infused at 800 pmol/kg/min for 180 minutes

Data and Safety Monitoring Plan: The DSMB will meet at least 3 times, once to review and ratify its charter, a second time to evaluate the safety data after 5 POTS patients finish the study, and every 6 months until year 5. These reports will provide information regarding recruiting, safety reporting, data quality, and efficacy. The committee will assess safety data including common adverse events, hospitalizations, and other serious adverse events.

Statistical Considerations: Standard graphing and screening techniques to detect outliers and to ensure data accuracy. The summary statistics for both continuous and categorical variables will be provided by subject groups for Aim 1. All hypotheses will be tested at the level of α=0.05. Open-source statistical package R (R Core Team, 2020) for analyses will be used.

For Aim 1, the primary endpoint is splanchnic venous capacitance (SVC). The comparison between POTS and HC groups on this endpoint will be made using either the two-sample t-test or the Wilcoxon Rank Sum test. Furthermore, this endpoint will be analyzed using the general linear model (GLM) with a set of covariates including age, body mass index in addition to the baseline measure of adjusted in the model. Other endpoints will be analyzed similarly as the primary endpoint.

Hemodynamic Parameters and Autonomic Measurements:

Hemodynamic data will be recorded using the WINDAQ data acquisition system (DI220, DATAQ, Akron, OH, 14 Bit, 1000Hz), and will be processed off-line using a custom written software in PV-Wave language (PV-wave, Visual Numerics Inc., Houston, TX). Detected beat-to-beat values of R-R intervals (RRI) and blood pressure will be interpolated and low-pass filtered (cutoff 2 Hz).

Data segments of at least 180 seconds will be used for spectral analysis. Linear trends will be removed, and power spectral density will be estimated with the FFT-based Welch algorithm. The total power (TP) and the power in the low (LF: 0.04 to <0.15 Hz), and high (HF: 0.15 to < 0.40 Hz) frequency ranges will be calculated . Cross spectra, coherence and transfer function analysis will be used to capture interrelationships between R-R interval and systolic blood pressure.

The baroreflex gain will be determined as the mean magnitude value of the transfer function in the low-frequency band, with a negative phase and squared coherence value greater than 0.5. Beat-to-beat stroke volume will be estimated by pulse contour analysis of arterial pressure curves (Modelflow algorithm) using a finger photo plethysmography volume-clamp BP device (Nexfin, BMEYE) and by impedance cardiography. An appropriate size cuff will be wrapped around the right middle or index finger and a height correction system will be used to adjust for hydrostatic height differences between the hand and the heart. Beat-to-beat BP data will be calibrated to brachial artery pressure and intermittently checked against oscillometric BP measurements (Dinamap ProCare, GE Healthcare). Then cardiac output will be calculated by multiplying stroke volume by the heart rate obtained from oscillometric BP measurements. Systemic vascular resistance will be estimated by dividing oscillometric mean arterial pressure (MAP) by cardiac output.

Superior Mesenteric Artery Flow Assessment: The superior mesenteric artery (SMA) flow will be studied using a sonographic system with real-time B-mode imaging coupled with pulsed Doppler and colour coded Doppler imaging (Philips EPIC 7C). Examination will be performed with a 3.5-Mhz phased array sector scanning probe (Philips C5-1 curved array transducer). The Doppler sample volume will be put about 2-cm downstream of the vessel's origin from the aorta. The peak systolic (S) and peak end-diastolic (D) Doppler frequencies will be measured on the time-frequency Doppler spectrum, and the resistance index (RI) will be calculated as: RI=(S-D)xS-1.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 50years of age
* Cases: Diagnosis of POTS with presyncope symptoms after meals Or

Controls:

* With no significant past medical history, non-smokers and not on chronic medications.
* Body mass index (BMI) between 18.5 to 29.9 kg/m2
* If pre-menopausal women: must have regular menstrual cycle.

Exclusion Criteria:

* BMI above ≥30 kg/m2
* Irregular menstrual cycle
* Intolerance to CPAP.
* Chronic use of acetaminophen
* Heart problems: myocardial infarction, angina, heart failure, stroke
* Undergone any heart related procedures or stents or on pacemaker.
* Uncontrolled hypertension.
* Type 1 or type 2 diabetes mellitus
* Pregnant or breast-feeding women.
* Impaired liver function
* Impaired Kidney function test.
* Anemia (Hematocrit<34%).
* Ongoing substance abuse.
* Subjects with abnormal EKG
* History of seizures.
* Diagnosed with neuropathy due to any reason
* History of neck surgery.
* Smoker,
* On statin therapy for high cholesterol
* Rheumatoid arthritis.
* On oral corticosteroids,
* Current infections
* Documented of moderate decrease in blood volume

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-25 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in splanchnic venous capacitance in Postural Orthostatic Tachycardia Syndrome | Baseline up to 180 minutes post glucose challenge
  The changes in splanchnic venous capacitance and superior mesenteric arterial flow will be measured, before and after a 75 gram of oral glucose challenge. It will compared in POTS and Healthy controls.
  While segmental bio impedance is monitored, continuous positive airway pressure (CPAP) will be applied sequentially at 0, 4, 8, 12 and 16 cm H2O for about 30 seconds each; this positive airway pressure will increase the intrathoracic pressure, which is transmitted to the venous circulation. Pressure (CPAP pressure, x-axis) - volume (splanchnic vascular volume measured by segmental impedance and expressed as % change from baseline, y-axis) relationships are then constructed to assess for splanchnic venous capacitance.
Effect of glucose-induced GIP secretion on splanchnic venous capacitance | 0-180 mins
  25 participants with POTS diagnosis, will be randomized them to either saline versus GIP antagonist (GIP(3-30)NH2) acute infusion. We will measure changes in their splanchnic venous capacitance and superior mesenteric arterial flow before and after a 75-g oral glucose challenge during supine and 45-degree head-up tilt positions (orthostatic challenge) for up to 3 hr
Effect of glucose-induced GIP secretion on POTS postprandial symptoms. | 0-90 mins
  Compare the post prandial symptoms on the participants who got infused with GIP antagonist GIP(3-30)NH2 and compare it with Saline infused participants at baseline and 45 degree head tilt. Total of 25 participants with diagnosis of POTS will randomized at visit 2, as 1:1 saline vs GIP antagonist GIP(3-30)NH2 At visit 3, the subjects who received Saline, will get GIP antagonist GIP(3-30)NH2 , vice versa.

SECONDARY OUTCOMES:
Measure Glucose-dependent Insulinotropic polypeptide (GIP) hormone level in POTS patients and Controls after 75 grams of glucose ingestion | Baseline up to 180 minutes post glucose challenge
  Measure and compare various GIP hormones (GLP-1, GLP-2, GIP, Vasoactive Intestinal Peptide(VIP)and glucagon) after ingesting 75-gram glucose for up to 180 minutes in POTS patients and healthy controls of similar age and BMI.
  Sequential blood draw will done to measure GIP hormones

CONTACTS AND LOCATIONS:
Overall Officials: Cyndya Shibao, M.D, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jacob G, Costa F, Shannon JR, Robertson RM, Wathen M, Stein M, Biaggioni I, Ertl A, Black B, Robertson D. The neuropathic postural tachycardia syndrome. N Engl J Med. 2000 Oct 5;343(14):1008-14. doi: 10.1056/NEJM200010053431404. PMID 11018167
- [Result] Shibao C, Arzubiaga C, Roberts LJ 2nd, Raj S, Black B, Harris P, Biaggioni I. Hyperadrenergic postural tachycardia syndrome in mast cell activation disorders. Hypertension. 2005 Mar;45(3):385-90. doi: 10.1161/01.HYP.0000158259.68614.40. Epub 2005 Feb 14. PMID 15710782
- [Result] Prentky RA, Watt NF, Fryer JH. Longitudinal social competence and adult psychiatric symptoms at first hospitalization. Schizophr Bull. 1979;5(2):306-12. doi: 10.1093/schbul/5.2.306. PMID 462143
- [Result] Bourne KM, Stiles LE, Raj SR, Shibao CA. Do meals affect heart rate and symptoms in postural orthostatic tachycardia syndrome? Clin Auton Res. 2022 Feb;32(1):65-67. doi: 10.1007/s10286-021-00835-0. Epub 2021 Nov 18. No abstract available. PMID 34792683
- [Result] Breier NC, Paranjape SY, Scudder S, Mehr SE, Diedrich A, Flynn CR, Okamoto LE, Hartmann B, Gasbjerg LS, Shibao CA. Worsening Postural Tachycardia Syndrome Is Associated With Increased Glucose-Dependent Insulinotropic Polypeptide Secretion. Hypertension. 2022 May;79(5):e89-e99. doi: 10.1161/HYPERTENSIONAHA.121.17852. Epub 2022 Mar 2. PMID 35232225